CLINICAL TRIAL: NCT00266097
Title: A Two-Part Phase I Study of the Addition of Oxaliplatin to Gemcitabine, and Then Erlotinib Plus Oxaliplatin to Gemcitabine as Radiosensitizers for Pancreatic and Biliary Adenocarcinoma
Brief Title: Oxaliplatin, Gemcitabine, Erlotinib, and Radiation Therapy in Treating Patients With Unresectable and/or Metastatic Pancreatic Cancer or Biliary Tract Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0405; P30CA016086 (NIH); CDR0000550061 (Other: PDQ number)
Record Dates: First submitted 2005-12-13; First posted 2005-12-15 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Extrahepatic Bile Duct Cancer; Gallbladder Cancer; Pancreatic Cancer
Keywords: stage III pancreatic cancer; stage IV pancreatic cancer; unresectable extrahepatic bile duct cancer; unresectable gallbladder cancer; adenocarcinoma of the extrahepatic bile duct; adenocarcinoma of the gallbladder; adenocarcinoma of the pancreas; recurrent pancreatic cancer; recurrent extrahepatic bile duct cancer; recurrent gallbladder cancer
MeSH Terms: conditions — Bile Duct Neoplasms; Gallbladder Neoplasms; Pancreatic Neoplasms | interventions — Erlotinib Hydrochloride; Gemcitabine; Oxaliplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part I (Experimental): Oxaliplatin + Gemcitabine + Radiation
  Interventions: Drug: gemcitabine hydrochloride; Drug: oxaliplatin; Radiation: radiation therapy
- Part II (Experimental): Erlotinib + Oxaliplatin + Gemcitabine + Radiation
  Interventions: Drug: erlotinib hydrochloride; Radiation: radiation therapy; Drug: gemcitabine hydrochloride; Drug: Oxaliplatin

INTERVENTIONS:
Drug: erlotinib hydrochloride — Cohort (-1) = 50 mg daily Cohort 1 = 50mg daily Cohort 2= 75 mg daily Cohort 3 = 100mg daily Cohort 4 = 100mg daily Cohort 5 = 150mg daily
  Arms: Part II
Drug: gemcitabine hydrochloride — Gemcitabine will be given at a dose of 100 mg/m2 for the first cohort and escalated to a fixed dose of 200 mg/m2 for the remaining 3 cohorts
  Arms: Part I
Drug: oxaliplatin — Oxaliplatin will be given at 30 mg/m2 weekly for the first two cohorts and then will be dose-escalated to 45 mg/m2 and 60 mg/m2 for the next 2 in cohorts
  Arms: Part I
Radiation: radiation therapy — 5040 cGy, every week, up to 6 weeks
Drug: gemcitabine hydrochloride — Given weekly at a starting dose of 100mg/m2 in the first 3 cohorts and dose escalated to 200 mg/m2 for the remaining 2 cohorts
  Arms: Part II
Drug: Oxaliplatin — The Part II dose of oxaliplatin will be determined by Part I of the study. The dose for Part II will be one dose level increase from the MTD determined in Part I.
  Arms: Part II

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin and gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving oxaliplatin together with gemcitabine, erlotinib, and radiation therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of oxaliplatin, gemcitabine, and erlotinib when given together with radiation therapy in treating patients with unresectable and/or metastatic pancreatic cancer or biliary tract cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose (MTD) of oxaliplatin and gemcitabine hydrochloride when combined with radiotherapy in patients with unresectable and/or metastatic pancreatic or biliary tract adenocarcinoma. (Part 1)
* Determine the MTD of erlotinib hydrochloride and gemcitabine hydrochloride when combined with oxaliplatin at the MTD and radiotherapy in these patients. (Part 2)

OUTLINE: This is a multicenter, nonrandomized, parallel group, uncontrolled, open-label, dose-escalation study of gemcitabine hydrochloride, oxaliplatin, and erlotinib hydrochloride.

* Part 1: Patients receive gemcitabine hydrochloride IV over 30-60 minutes and oxaliplatin IV on day 1. Patients also undergo external beam radiotherapy (EBRT) once daily on days 1-5. Treatment repeats every 7 days for up to 6 courses.

Cohorts of 3-6 patients receive escalating doses of gemcitabine hydrochloride and oxaliplatin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity (DLT). Up to 10 patients are treated at the MTD.

* Part 2: Patients receive gemcitabine hydrochloride, oxaliplatin*, and EBRT as in part 1. Patients also receive oral erlotinib hydrochloride once daily on days 1-5. Treatment repeats every 7 days for up to 6 courses.

Cohorts of 3-6 patients receive escalating doses of gemcitabine hydrochloride and erlotinib hydrochloride until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience DLT. Up to 10 patients are treated at the MTD.

NOTE: *Patients receive oxaliplatin at the MTD determined in part 1.

After completion of study treatment, patients are followed every 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy confirmed diagnosis of any of the following:

  * Pancreatic carcinoma
  * Ampullary carcinoma
  * Biliary tract (gallbladder or bile duct) carcinoma
* Unresectable and/or biopsy-proven metastatic disease
* Suitable for bimodality therapy, as determined by a medical oncologist and radiation oncologist

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 2 months
* ANC > 1,500/mm³
* Platelet count > 100,000/mm³
* Creatinine < 1.5 mg/dL
* Total bilirubin < 2 times upper limit of normal (ULN)
* AST < 3 times ULN (< 5 times ULN if liver metastases are present)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known hypersensitivity to platinum agent or gemcitabine hydrochloride
* No serious medical or psychiatric illnesses that would preclude giving informed consent

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy to the upper abdomen
* More than 3 weeks since prior chemotherapy
* No prior erlotinib hydrochloride
* At least 5 days since prior and no concurrent CYP3A4 inducer/inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2004-08; Primary Completion 2009-03 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of oxaliplatin and gemcitabine hydrochloride (Part 1) | 6 weeks
  The MTC of Oxaliplatin and gemcitabine is defined as the combination for which the rate of toxicities that cause dose reductions plus twice the rate of dsoe limiting toxicity (DLT) is equal to 0.5
Maximum Tolerated Dose (MTD) of erlotinib hydrochloride and gemcitabine hydrochloride (Part 2) | 6 weeks
  The highest dose for which the observed dose reduction rate plus twice the dose limiting toxicity (DLT) rate does not exceed 0.5 will be declared the MTD

CONTACTS AND LOCATIONS:
Overall Officials: Bert H. O'Neil, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States